CLINICAL TRIAL: NCT05088928
Title: Efficacy and Safety of Apixaban in COVID-19 Coagulopathy Patients With Respiratory Severity Under Critical
Brief Title: Efficacy and Safety of Apixaban in COVID-19 Coagulopathy Patients With Respiratory Severity Under Critical Care
Acronym: ECRU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Scotmann Pharmaceuticals (Industry)
Collaborators: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Dr. Syeda Saba Aslam, Head of Medical Affairs, Scotmann Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMUSCOTMANNECRUTRIAL; U1111-1272-7249 (Registry Identifier: ICTRP, WHO)
Record Dates: First submitted 2021-10-21; First posted 2021-10-22 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: Anticoagulation; Apixaban
MeSH Terms: conditions — COVID-19 | interventions — apixaban; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Experimental): Ecru (Apixaban )Tablets
  Interventions: Drug: Apixaban
- Comparator/control (Active Comparator): Rivascot (Rivaroxaban)
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Apixaban — Direct Acting Oral Anti coagulant
  Other Names: ECRU Tablets
  Arms: Interventional Arm
Drug: Rivaroxaban — Direct Acting Oral Anti coagulant
  Other Names: Rivascot tablets
  Arms: Comparator/control

SUMMARY:
The purpose of the study is to describe the safety and efficacy outcomes of a cohort of ICU patients with severe COVID-19 respiratory disease treated with therapeutic dose Apixaban for COVID-19 at a tertiary public health care setting.

DETAILED DESCRIPTION:
There is an increased risk of Venous and Arterial thromboembolism in COVID-19 infection. The main reason being that the novel coronavirus SARS-CoV-2 induces hyperinflammation and subsequently immunothrombolism which is wide spread in the body. The angiotensin converting enzyme 2 (ACE2) receptor, which is utilized by the virus to infect the host, is present throughout the human body organs and endothelial cells. Thrombotic microangiopathies are the consequence of this direct endothelial invasion of the virus and widespread endothelial inflammation. Consequently, pervasive dysfunction of the endothelium and apoptosis is seen primarily due to the host immune response and release of pro inflammatory cytokines.

A hypercoagulable state is therefore seen due to the shift in the vascular equilibrium towards a vasoconstrictive and inflammatory response, promoting a microvascular derangement and dysfunctions.

Although this pathological response is not unique to the COVID-19 disease, the systemic coagulopathies observed due to this novel virus are noted to be slightly distinct. These include the increased risk of mortality with the increased level of D-Dimers in nearly 50% of the patients . While mild prolongation of Prothrombin time and thrombocytopenia are not noted to be important predictors of the severity of the disease or its adverse outcomes .

In COVID-19 patients, the International Society on Thrombosis and Hemostasis (ISTH). criteria for Disseminated Intravascular Coagulation (DIC) is seldom met, despite the indication by the typical triad of thrombin time prolonged, decreased platelet counts and increased D-dimer levels .

Although the Disseminated Intravascular Coagulation is low grade, the fibrinolytic system is activated and endogenous tissue plasminogen is released because of the pathogenic inflammation-causing endothelial cell injury and thrombotic angiopathies of the microvascular system. This also contributes to the increased mortalities due to high D-Dimer levels.

WHAT IS KNOWN?

As high as 69% of COVID-19 patients under Critical Care have been reported to experience the incidence of complication related to thromboembolism .

Although the use of unfractionated heparin (UFH) or low molecular weight heparin (LMWH) as anticoagulation prophylaxis has been observed with beneficial results in decreasing COVID-19 mortalities, however, there are reports of high incidences of thromboembolic complications despite the prophylaxis too.

Although prophylactic therapeutic anti coagulation has been reported with reduced incidences of venous thromboembolism (VTE) , a study has shown almost similar incidence of bleeding in the anticoagulation prophylaxis group as compared to the group which did not receive any anticoagulation (3 versus 1.9%, p = 0.20).

RATIONALE:

Since the link between COVID-19 related coagulopathies and mortalities has been established, it is of paramount importance to establish the optimal strategy. When compared to classical anticoagulants including Unfractioned Heparin, the comparatively newer salt of Apixaban belonging to the Direct Oral Anti Coagulants (DOACs) class, has been reported to have decreased rate of unwanted bleeding incidences, lower requirement of regular lab monitoring, fewer drug-drug interactions, increased pharmacokinetic (PK) and pharmacodynamic (PD) predictability and better efficacy .

Due to these advantages particularly the more predictable dose-response curve of Apixaban, its use has markedly increased in many generalized settings in hospitals since its approval. Apart from this, it is also being started in the Critical Units of COVID-19 and continued thereafter.

RELEVANCE, IMPORTANCE AND APPLICABILITY:

The investigators had particular interest in Apixaban in the COVID-19 setting because of the easy twice daily dosing regime, decreased need of regular lab monitoring, decreased room congestion, decreased medical staff exposure and consequently decreased need of Personal Protective Equipment among others. Nevertheless, the anti-inflammatory effects of Apixaban by decreasing plasma induced superoxide productions, are comparable to Unfractioned Heparin and Low Molecular Weight Heparin.

RESEARCH GAP IDENTIFIED:

Despite these numerous purported benefits, to the best of the investigators' knowledge, there are no published reports describing the clinical outcomes of apixaban use in critically ill ICU patients with severe COVID-19 , in Pakistan.

PURPOSE OF STUDY:

As such, the purpose of this study is to describe the safety and efficacy outcomes of a cohort of ICU patients with severe COVID-19 respiratory disease treated with therapeutic dose apixaban for COVID-19 at a tertiary public health care setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age)
* All admitted patients with severe or critical COVID-19
* Confirmed diagnosis of COVID-19 through RT-PCR (attach report) and/or HRCT Chest
* Patients at high risk of coagulopathy demonstrating signs of micro-thrombi induced organ dysfunction or strongly suspected macro thromboembolism

Exclusion Criteria:

* High risk of bleeding as judged by treating physicians
* Contra-indication to therapeutic anti coagulation
* Platelets < 50,000 (attach report)
* INR >1.5
* Evidence of current or recent bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding | 10 days
  The participants with bleeding episodes

SECONDARY OUTCOMES:
Clotting | 10 days
  The participants with clotting incidences

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muhammad Umar, MBBS, Principal Investigator — Rawalpindi Medical College
Locations (1):
- Rawalpindi Medical University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Proformas